CLINICAL TRIAL: NCT00382798
Title: A Multiple-Center, Observer-Blinded, Randomized, Placebo-Controlled, Single & Multiple Ascending Dose Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, & Food Effect of RO5024048 in Healthy Volunteers & in Patients With Chronic HCV Infection
Brief Title: Adaptive Phase I HCV Study With Nucleoside Analogue, in Combination With Interferon and Ribavirin
Acronym: R7128
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmasset (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Amanda Beard, Pharmasset, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P7081-5101
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Volunteers; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: RO5024048

SUMMARY:
This is an adaptive Phase I study to evaluate RO5024048 in the following groups:

* Healthy Volunteers (Part 1 - Single Ascending Dose Study) -Enrollment completed
* Hepatitis C virus (HCV) genotype 1 infected patients who have failed interferon therapy (Part 2- Multiple Ascending Dose Study)-Enrollment Completed
* HCV genotype 1-infected patients who are treatment naive, to be dosed in combination with PEG-IFN and RBV (Part 3 - Combination Dose Study)-Currently Enrolling
* HCV genotype 2-3 infected patients who have previously been treated with interferon but who did not respond, to be dosed in combination with PEG-IFN and RBV (Part 3 - Combination Dose Study)- Currently enrolling

The study aims to determine if RO5024048 is safe and well-tolerated in healthy people and in people infected with hepatitis C virus. The amount of RO5024048 in the blood will be measured during the study and the amount of hepatitis C virus in the blood after each dose will also be measured.

During Part 3 of the study, RO5024048 will be given with PEG-IFN and RBV, two drugs currently used and approved for the treatment of HCV.

DETAILED DESCRIPTION:
Part 3: During Part 3 of the study, HCV gentoype 1-infected patients who are treatment-naive (have not been treated for HCV) will be enrolled. Up to 75 patients (3 groups of 25) will be dosed for 28 days with RO5024048, PEG-IFN, and RBV. The first dose of RO5024048 to be given in Part 3 will be 500 mg BID, the second dose will be 1500 mg BID, and the third group will be 1000 mg BID. Standard doses of PEG-IFN and RBV will be used during Part 3. Doses of PEG-IFN and RBV will be modified if necessary.

An 4th group of 25 HCV genotype 2 or 3-infected patients who have been previously treated with interferon but who did not respond will also be enrolle in part 3. The dose given to this 4th group will be 1500 mg BID, in combination with standard doses of PEG-IFN and RBV.

Following 28 days of combination dosing with RO5024048, PEG-IFN, and RBV, patients will be dosed an additional 28 days (through Day 56 of the study) with just PEG-IFN, and RBV. After completing 56 days under this study, patients who participate in Part 3 will be optionally enrolled into a standard of care protocol with PEG-IFN and RBV, to be conducted by Roche. Patients who opt to enroll into the standard of care protocol will be given up to 40 weeks of PEG-IFN and RBV.

The primary objective for Part 3 is to assess the safety, tolerability and pharmacokinetics of RO5024048 in treatment-naive HCV Genotype 1-infected patients, and in non-responder HCV Genotype 2/3-infected patients, after once or twice daily dosing in combination wtih PEG-IFN and RBV for 28 days on an outpatient basis. The secondary objective of Part 3 (COMBO) is to evaluate the short-term decrease in viral load in treatment-naive HCV Genotype 1-infected patients, and in non-responder HCV Genotype 2/3-infected patients, after once or twice daily dosing of RO5024048 in combination with PEG-IFN and RBV for 28 days.

Part 1 (closed for enrollment): Single ascending dose study

During Part 1, 5 escalating single oral doses of RO5024048 or placebo were given to 40 healthy volunteers, when fasted (have not eaten any food for at least 10 hours). The doses given were 500 mg, 1500 mg, 4500 mg, 6000 mg, and 9000 mg. Another group of 6 volunteers was given 1500 mg with food.

The primary objective of Part 1 was to assess the safety, tolerability, and pharmacokinetics (amount of drug in the blood) of RO5024048 under fasting conditions. The secondary objective of Part 1 was to explore the effect of food on the pharmacokinetics of RO5024048.

Part 2: (Closed for enrollment) Multiple ascending dose study

During Part 2 of the study, 40 HCV-genotype 1-infected patients were given multiple-ascending oral doses of RO5024048 or placebo for 14 days. The doses given were 750 mg once daily, 1500 mg once daily, 750 mg twice daily, and 1500 mg twice daily.

The primary objective of Part 2 was to assess the safety, tolerability and pharmacokinetics of RO5024048 in HCV Genotype 1-infected patients after daily or twice daily dosing for 14 days. The secondary objective was to evaluate the decrease in viral load in HCV Genotype 1-infected patients after daily or twice daily dosing of RO5024048 for 14 days

ELIGIBILITY:
Inclusion Criteria Part 3:

* Males or females of non-childbearing potential aged 18 to 65 years. Females must be surgically sterile, or post-menopausal for at least 12 months. Females of child-bearing potential may be enrolled provided they use two methods of acceptable contraception.
* Diagnosed with chronic liver disease consistent with chronic hepatitis C infection, genotype-1, for at least 6 months.
* Genotype 1 Patients who are HCV treatment-naive, with no history of exposure to interferon, ribavirin, or direct antivirals; OR Genoytpe 2 or 3 patients who have previously been treated with interferon.
* Otherwise healthy as determined at screening.
* At least one measurement of serum HCV RNA of ≥ 100,000 IU/mL measured during Screening by the COBAS AmpliPrep/COBAS TaqMan HCV.
* ALT and AST measurement at Screening < 5 times of ULN.
* Liver biopsy obtained within 2 years (24 calendar months) prior to Screening with a fibrosis classification of non-cirrhotic as judged by a local pathologist. Incomplete cirrhosis (Ishak 5) is also considered as cirrhosis. If no history of liver biopsy, a study qualifying biopsy must be performed during the screening period, prior to randomization.
* Negative pregnancy test (for all females) at Screening and Day -1.
* All male patients with female partners of child-bearing potential must use two acceptable methods of contraception (one of which must be a barrier method), during and for 3 months after participation in the study.
* A body mass index (BMI) of ≥ 18 kg/m2, but not exceeding 36.
* Able to abstain from any alcohol (including alcohol-containing products) and able to limit caffeine consumption to two 8-ounce cups of coffee or the equivalent per day, from 72 hours before receiving study drug through the end of the study (Day 56 or early termination).
* Able to effectively communicate with the Investigator and other testing center personnel.
* Able to participate and willing to give written informed consent and comply with the study restrictions.

Exclusion Criteria

* Positive test at Screening for HAV, HBV, or HIV.
* History or other evidence of a medical condition associated with chronic liver disease, decompensated liver disease, renal disease, immunologically mediated disease, chronic pulmonary disease, cardiac disease, thyroid disease, severe retinopathy, severe psychiatric disease, organ transplantation, cancer, seizure disorder, or pancreatitis.
* Abnormal hematological, biochemical, or coagulation parameters at Screening; or positive fecal occult blood test.
* Estimated creatinine clearance of 90 mL/minute or less at Screening.
* Poorly controlled hypertension, or anyone who at screening or baseline has a BP of 140/90 or greater.
* Type 1 or 2 diabetics with hemoglobin A1C > 7.
* A baseline increased risk for anemia.
* Screening ECG QTc value ≥ 450 ms and/or clinically significant ECG findings.
* Positive results for drugs of abuse at Screening.
* History of clinically significant drug allergy to nucleoside/nucleotide analogues.
* Donation or loss of more than 400 mL blood within 2 months prior to anticipated dose administration.
* Participation in a clinical study with an investigational drug, biologic, or device within 3 months prior to anticipated dose administration.
* Males whose female partner is pregnant.
* Any chronic viral (including HSV), bacterial, mycobacterial, fungal, parasitic, or protozoal infection.
* Serum alpha-feto-protein > 50 ng/mL at screening.
* Receipt of any vaccination within 30 days prior to anticipated dose administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Michelle Berrey, MD, Study Director — Pharmasset
Locations (9):
- United States (7):
  - Quest Clinical Research, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Duke Clinical Research Institute, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Auckland Clinical Studies Limited, Grafton, Auckland, New Zealand
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico